CLINICAL TRIAL: NCT07340281
Title: Examining Novel Biomarkers of Neuroplasticity Associated With Exercise in Adults With Anxiety Disorders
Brief Title: Biomarkers for Exercise
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 25-01561
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individuals with Anxiety Disorder (Experimental): All participants will complete the 4-week exercise intervention in which they'll be prescribed 150 minutes of moderate intensity exercise per week at home, which will be measured using Fitbits.
  Interventions: Behavioral: Exercise Intervention
- Control Individuals (Active Comparator): All participants will complete the 4-week exercise intervention in which they'll be prescribed 150 minutes of moderate intensity exercise per week at home, which will be measured using Fitbits.
  Interventions: Behavioral: Exercise Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — Exercise intervention is delivered in weekly individual sessions virtually for the 4-week intervention period. Sessions range from 25-45 minutes. The sessions serve as touch base points to review exercise for the week, plan for the coming week, problem-solve obstacles, and discuss various motivational strategies to help with an exercise routine. Participants are prescribed 150 minutes of moderate intensity exercise per week to be completed at home.

SUMMARY:
The overarching objective is to examine the brain-based biological mechanistic pathway by which exercise exerts anxiolytic effects. The investigators will measure brain-derived markers of mitochondrial metabolism (acetyl-L-carnitine [LAC]) and inflammation (interleukin-6 [IL-6]) using innovative technology to isolate neuronal exosomes.

ELIGIBILITY:
Inclusion Criteria:

For both participant groups: To be eligible to participate in this study, an individual must meet all of the following criteria:

* Between 18-50 years of age
* Currently sedentary (≤60 minutes of moderate intensity exercise per week for the past 3 months)
* Capable and willing to provide informed consent

For anxiety disorder participant group, an individual must also meet:

• Primary psychiatric diagnosis of generalized anxiety disorder (GAD), social anxiety disorder, or panic disorder

Exclusion Criteria:

* Lifetime history of Bipolar I or II or any psychotic disorder
* Bulimia or anorexia in the past 3 months
* Alcohol or substance use disorder in the past 3 months
* Current major depressive disorder (past is allowed)
* Current neurologic disorder
* High current suicide risk (active suicidal ideation with plan and intent) as indicated by a score of ≥4 on the Columbia Suicide Severity Rating Scale (C-SSRS) consistent with a need for referral to higher level of care
* Participation in concurrent evidence-based therapy (e.g., cognitive behavioral therapy) targeting anxiety and/or depression (supportive therapy and couples therapy are allowed)
* Risk for exercise according to the Physical Activity Readiness Questionnaire with excluded active medical conditions including heart conditions, lung disease, bone/joint problems, or seizures
* Women who are currently pregnant or plan to become pregnant during the duration of the study
* current psychiatric medication
* Current substance abuse or positive urine toxicology screen (recreational use of marijuana is permitted based on clinical assessment on the MINI structured diagnostic interview that it does not meet criteria for cannabis use disorder)
* Active infection

Non-psychiatric controls who meet the following criteria will be excluded from participation in this study:

• Current psychiatric condition assessed by the MINI

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Acetyl-L-carnitine (LAC) Levels | Week 4
  Levels of LAC isolated from neuronal exosomes from plasma blood draws.
Interleukin-6 (IL-6) Levels | Week 4
  Levels of IL-6 isolated from neuronal exosomes from plasma blood draws.

SECONDARY OUTCOMES:
Continuously measured moderate/vigorous minutes of exercise | Up to Week 4
  Information collected via Fitbit.
7-Day Physical Activity Recall | Baseline, Week 2, Week 4
  Measurement of total weekly metabolic equivalent of task (MET)-hours.
Overall Anxiety Severity and Impairment Scale (OASIS) | Baseline, Week 2, Week 4
  OASIS is a 5-item assessment of anxiety severity and impairment over the past week; each item is rated on a Likert scale from 0-4. The total score is the sum of responses and ranges from 0-20; higher scores indicate greater anxiety severity and impairment.
Anxiety Sensitivity Index (ASI-3) Score | Baseline, Week 2, Week 4
  ASI-3 is an 18-item assessment of anxiety severity over the past week; each item is rated on a Likert scale from 0-4. The total score is the sum of responses and ranges from 0-72; higher scores indicate greater anxiety severity.
Quick Inventory of Depressive Symptomatology (QIDS) Score | Baseline, Week 2, Week 4
  QIDS is a 16-item assessment of depressive symptomatology; each item is rated on a Likert scale from 0-3. The total score is the sum of responses from each of the 9 domains and ranges from 0-27; higher scores indicate greater severity of depressive symptomatology.
Perceived Stress Scale (PSS) Score | Baseline, Week 2, Week 4
  PSS is a 10-item assessment of perceived stress; each item is rated on a scale from 0-4. The score is the sum of responses ranges from 0 to 40 with higher scores indicating higher perceived stress.
Childhood Trauma Questionnaire | Baseline, Week 2, Week 4
  CTQ is a 28-item assessment of childhood trauma. The scale comprises five sub-scales; the score to each subscale ranges from 5-25; the total score is the sum of the sub-scales and ranges from 25-125; higher scores indicate more frequent/severe childhood trauma experiences.
Insomnia Severity Index (ISI) Score | Baseline, Week 2, Week 4
  ISI is a 7-item assessment of insomnia; each item is rated on a scale from 0-4. The total score is the sum of responses and ranges from 0-28; higher scores indicate greater insomnia severity.
International Physical Activity Questionnaire (IPAQ) Score | Baseline, Week 2, Week 4
  IPAQ is an assessment of overall activity levels; the total score is expressed as METs (Metabolic Equivalents), a unit representing energy cost, where 1 MET is resting energy expenditure.
Body Mass Index (BMI) | Baseline, Week 2, Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Szuhany, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data will be made available if requested.